CLINICAL TRIAL: NCT04630665
Title: Clinical Assessment of Buccal Bone Resorption in Immediate Implants in Thin and Thick Buccal Plates of Bone and Its Implication on Esthetics. A Controlled Clinical Trial
Brief Title: Buccal Bone Resorption in Immediate Implants in Thin and Thick Buccal Plates of Bone in Esthetic Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzy Nabil Naiem, Principal Investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21 Dec 2018 Protocol
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Buccal Bone Thickness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thin buccal bone (Other): immediate implant placement in thin buccal bone wall socket
  Interventions: Other: immediate implant placement
- ≥1 buccal bone (Other): immediate implant placement in 1 mm or more buccal bone thickness socket
  Interventions: Other: immediate implant placement

INTERVENTIONS:
Other: immediate implant placement — immediate implant placement in thin and thick buccal bony plates

SUMMARY:
To achieve esthetic immediate implants a minimum of adequate buccal bone thickness must be present. It was postulated that 2 mm of buccal bone thickness was needed to prevent recession of the buccal plate. However, this was reduced to 1 mm with more ongoing research. In a recent study postulated that a buccal bone thickness less than 1 mm could be sufficient.

Scarce literature was found that monitored the ridge alterations following implant placement.

In regards to the controversies regarding the minimal initial buccal bone thickness required to perform immediate implant placement, our study aims to monitor the buccal bone thickness and soft tissue changes over a year from implant and prosthetic placement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have at least one unrestorable tooth in the esthetic zone that needs to be extracted.
* Subjects with healthy systemic condition.
* Availability of bone apical and palatal to the socket to provide primary stability.

Exclusion Criteria:

* Patients with signs of acute infection related to the area of interest.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits.
* Smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
buccal bone thickness | 1 year
  measurement of buccal bone thickness by a specially designed device and cone-beam computed tomography (CBCT) analysis

SECONDARY OUTCOMES:
pink esthetic score (PES) | 1 year
  to assess esthetics, the score is from 0-14 0 being worst , 14 being best.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF
Time Frame: 6 months following publishing

REFERENCES:
- [Background] Merheb J, Vercruyssen M, Coucke W, Beckers L, Teughels W, Quirynen M. The fate of buccal bone around dental implants. A 12-month postloading follow-up study. Clin Oral Implants Res. 2017 Jan;28(1):103-108. doi: 10.1111/clr.12767. Epub 2016 Jan 8. PMID 26749417
- [Background] El Nahass H, N Naiem S. Analysis of the dimensions of the labial bone wall in the anterior maxilla: a cone-beam computed tomography study. Clin Oral Implants Res. 2015 Apr;26(4):e57-e61. doi: 10.1111/clr.12332. Epub 2014 Jan 23. PMID 24450845